CLINICAL TRIAL: NCT02657681
Title: Prevention of Levodopa-induced Dyskinesias by Transcranial Static Magnetic Field Stimulation (tSMS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación de investigación HM (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other); Hospital Nacional de Parapléjicos de Toledo (Other); Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Guglielmo Foffani, Principal Investigator, Fundación de investigación HM
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MJFOX-9205; 9205 (Other Grant/Funding Number: Michael J. Fox Foundation)
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Dyskinesia, Medication-Induced; Parkinson's Disease
MeSH Terms: conditions — Dyskinesia, Drug-Induced; Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- tSMS (Experimental): 30 min of tSMS, one session per day, for 9 days over 2 weeks
  Interventions: Device: tSMS
- sham (Placebo Comparator): 30 min of sham, one session per day, for 9 days over 2 weeks
  Interventions: Device: sham

INTERVENTIONS:
Device: tSMS — Transcranial static magnetic field stimulation (tSMS) is a non-invasive brain stimulation (NIBS) technique that decreases cortical excitability. Static magnetic fields suitable for tSMS are obtained with commercially available neodymium magnets. We will use a cylindrical neodymium magnet of 45 mm diameter and 30 mm of thickness, with a weight of 360 g (MAG45r; Neurek SL, Toledo, Spain), which will be applied with south polarity to the motor cortex, over the representational field of hand area contralateral to the more affected side of the body.
  Other Names: MAGmv1.0 with MAG45r, Neurek S.L. (Toledo, Spain)
  Arms: tSMS
Device: sham — A non-magnetic metal cylinder, with the same size, weight and appearance of the magnet, will be used for sham stimulation (MAG45s; Neurek SL, Toledo, Spain).
  Other Names: MAGmv1.0 with MAG45s, Neurek S.L. (Toledo, Spain)
  Arms: sham

SUMMARY:
This is a randomized sham-controlled double-blind study to test the hypothesis that transcranial static magnetic field stimulation (tSMS) of the motor cortex improves levodopa-induced dyskinesias in patients with Parkinson's disease. Half of the patients will receive real tSMS treatment, the other half will receive sham treatment (placebo).

ELIGIBILITY:
Inclusion Criteria:

* advanced idiopathic Parkinson's disease (Brain Bank criteria)
* optimal clinical response to dopaminergic medication (>30% UPDRS-III improvement)
* presence of clinically relevant levodopa-induced peak-dose dyskinesias in at least one upper limb

Exclusion Criteria:

* MRI-incompatible metal objects in the body (e.g. cardiac pacemakers)
* other main neuropsychiatric co-morbidity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the maximal dyskinesia severity within 90min after levodopa intake, as measured by objective evaluation with the Unified Dyskinesia Rating Scale (UDysRS) one day after the end of treatment. | One day after the end of treatment compared to baseline

SECONDARY OUTCOMES:
Change from baseline of the maximal dyskinesia severity within 90min after levodopa intake, as measured by objective evaluation with the Unified Dyskinesia Rating Scale (UDysRS) one week after the end of treatment. | One week after the end of treatment compared to baseline
Dyskinesia severity evaluated for each body segment | Baseline, one day and one week after the end of treatment
Subjective evaluation of the treatment, as measured by the patient global impression of change (PGIC) | One day and one week after the end of treatment
Change from baseline in motor symptoms, as measured by the MDS-UDPRS III scale | Baseline, one day and one week after the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Guglielmo Foffani, PhD, Principal Investigator — CINAC, Hospital Universitario HM Puerta del Sur
Locations (1):
- CINAC, Hospital Universitario Puerta del Sur, Móstoles, Madrid, Spain